CLINICAL TRIAL: NCT05647811
Title: A Phase Ib, Open Label, Dose Escalation Study of NM8074 in Subjects with C3 Glomerulopathy (C3G)
Brief Title: Study of NM8074 in Adult C3 Glomerulopathy Patients
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NovelMed Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NM8074-C3G-101
Record Dates: First submitted 2022-11-18; First posted 2022-12-13 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: C3 Glomerulopathy

STUDY DESIGN:
Intervention Model Description: The study will enroll a planned number of 18 patients as subjects for the trial with the potential for more enrollment. Each cohort will consist of 6 subjects in a total of three cohorts at doses of 5, 10, or 20 mg/kg NM8074. No more than two to three subjects will be dosed in a single day. Safety data will be assessed and reviewed by the Sponsor and Study Investigators for dosed subjects prior to dose escalation or dosing of the rest of the study subjects within the Cohort. Dose escalation will occur only after four (4) subjects have been dosed and safety data has been evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): 6 subjects will receive NM8074 at 5 mg/kg weekly.
  Interventions: Drug: NM8074
- Cohort 2 (Experimental): 6 subjects will receive NM8074 at 10 mg/kg every 2 weeks.
  Interventions: Drug: NM8074
- Cohort 3 (Experimental): 6 subjects will receive NM8074 at 20 mg/kg every 2 weeks.
  Interventions: Drug: NM8074

INTERVENTIONS:
Drug: NM8074 — NM8074 will be administered as an intravenous infusion. Multiple dosing duration will range from 5 to 9 weeks.

SUMMARY:
This is a Phase Ib, open-label, dose-escalation study designed to evaluate the safety, efficacy, and immunogenicity of NM8074 administered intravenously to patients with C3 Glomerulopathy.

DETAILED DESCRIPTION:
The proposed study, NM8074-C3G-101, will enroll a planned number of 18 patients, with the potential to enroll more patients. There will be 3 cohorts with 6 patients each dosed at 5, 10, or 20 mg/kg depending on which cohort they are assigned to. Enrollment in the subsequent higher dose level cohort will occur after the previous cohort has been evaluated for safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 and ≤ 65 years at the time of consent
* Diagnosis of C3 Glomerulopathy as confirmed by C3 nephropathy in biopsy within 12 months prior to enrollment
* Reduced serum C3 levels (defined as less than 0.85 x lower limit of the central laboratory normal range) at Screening
* Patients with confirmed proteinuria
* Willing and able to understand and complete informed consent procedures, including signing and dating the informed consent form (ICF), and comply with the study visit schedule
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must have a negative pregnancy test at screening and must agree to use highly effective methods of contraception during dosing and for 1 week after stopping of investigational drug
* Males must agree to use contraceptives and refrain from donating sperm for the duration of the study
* Patients must have documentation of previous vaccination or be willing to be vaccinated prior to dosing with NM8074. All patients will be vaccinated against Neisseria meningitidis, Streptococcus pneumoniae and Haemophilus influenzae according to the most current Advisory Committee on Immunization Practices (ACIP) recommendations.
* Estimated glomerular filtration (eGFR) rate of ≤ 60 ml/min but ≥ 20 ml/min

Exclusion Criteria:

* Use of other investigational drugs at the time of enrollment
* Patients with other renal diseases that would interfere with interpretation of the study
* Estimated glomerular filtration rate of ≤ 20 mL/min/1.73m2 based on Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) at Screening
* Has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times the upper limit of normal (xULN)
* Has a known history of meningococcal disease or N. meningitidis
* Currently active systemic infection or suspicion of active bacterial, viral, or fungal infection that requires antibiotic, antifungal, antiparasitic, or antiviral mediations
* Temperature > 38°C for more than two weeks prior to screening
* History of renal organ transplantation
* Pregnant, planning to become pregnant, or nursing female subjects
* C3G patients currently under complement blocker treatments
* Participation in any experimental small molecule or non-antibody therapy within 60 days prior to dosing on Day 1 (participation in observational studies and/or registry studies is permitted)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Monitoring for incidence of Adverse Events (AEs)/Serious Adverse Events (SAEs) | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
Change from Baseline or Percent Change from Baseline in Urine Protein to Creatine Concentration Ratio (UPCR) | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
Change from Baseline or Percent Change from Baseline in Urine Albumin to Creatinine Concentration Ratio (UACR) | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
Ratio to Baseline of UPCR and UACR | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
  Derived from 24h urine collection
Change from Baseline or Percent Change from Baseline in Estimated Glomerular Filtration Rate (eGFR) | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3

SECONDARY OUTCOMES:
Percent Change from Baseline in Alternative Pathway (AP) of Complement Activity as Compared to Percent Change from Baseline in Classical Pathway (CP) of Complement Activity as Measured by Percent Change in Levels of Membrane Attack Complex (MAC) | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
Percent Change from Baseline in Alternative Pathway (AP) of Complement Activity as Compared to Percent Change from Baseline in Classical Pathway (CP) of Complement Activity as Measured by Percent Change in Levels of Complement Component C3b | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
Change from Baseline or Percent Change from Baseline in Serum C3 Levels | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
Change from Baseline or Percent Change from Baseline in Glomerular Inflammation | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
  Measured by change from baseline or percent change from baseline in the C3G Histologic Index for Disease Activity - Combined C5b-9 Strata. Scores range from 0-21 where a decrease in score indicates improvement.
Change from Baseline or Percent Change from Baseline in Quality of Life (QoL) Assessed via the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale, Version 4. | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
  The FACIT-fatigue scale is a 13-item patient-reported measure of fatigue with a 7-day recall period. Items are scored on a 0 - 4 response scale ranging from "Not at all" to "Very much so". All items are summed to create a single fatigue score with a range from 0 to 52 with a better quality of life indicated by a higher score.
Change from Baseline or Percent Change from Baseline in Quality of Life (QoL) Assessed via the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 Scale (QLQ- C30), Version 3.0 | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
  All EORTC QLQ-C30 scales and single-item measures range from 0 to 100. This includes 3 symptom scales (fatigue, pain, nausea and vomiting), 5 functional scales (physical, role, cognitive, emotional, and social), single-item questions addressing symptoms like insomnia, dyspnea, loss of appetite, and others that are commonly reported by cancer patients, and the perceived financial impact of the disease. A higher score is associated with a greater quality of life for global health status.
Changes in plasma concentration of NM8074 | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
Maximum plasma concentration (Cmax) | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
Time corresponding to Cmax (tmax) | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
Area under the drug concentration-time curves (AUC0-t) | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
Change from Baseline or Percent Change from Baseline in Levels of Complement Component C3b via Alternative Pathway (AP) of Complement Activity | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
Change from Baseline or Percent Change from Baseline in Levels of Membrane Attack Complex (MAC) via Alternative Pathway (AP) of Complement Activity | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3

OTHER OUTCOMES:
Change from Baseline or Percent Change from Baseline in Levels of Complement Component C3b via Classical Pathway (CP) of Complement Activity. | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3
Change from Baseline or Percent Change from Baseline in Levels of Membrane Attack Complex (MAC) via Classical Pathway (CP) of Complement Activity. | Up to Study Day 50 for Cohort 1 and up to study day 84 for Cohort 2 and 3

IPD SHARING:
Plan to Share IPD: No